CLINICAL TRIAL: NCT06689345
Title: Effects of Non-invasive Neuromodulation on Post-COVID-19 Syndrome: Multicenter Study
Brief Title: Effect of Non-Invasive Neuromodulation on Primary Chronic Pain, Including Post-COVID-19
Status: Enrolling by invitation | Phase: Not Applicable | Type: Interventional
Sponsor: Federal University of ABC (Other)
Collaborators: University of Sao Paulo (Other); Coordination for the Improvement of Higher Education Personnel (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Sequential | Masking: Double | Purpose: Treatment
Other Study IDs: U1111-1293-2751
Record Dates: First submitted 2024-09-27; First posted 2024-11-14 (Actual); Last update posted 2024-11-14 (Actual); Status verified 2024-09

CONDITIONS: Post COVID Condition; Chronic Pain; Healthy
Keywords: neuromodulation; chronic pain; covid-19; TMS-EEG; vagal nerve
MeSH Terms: conditions — Post-Acute COVID-19 Syndrome; Chronic Pain; COVID-19

STUDY DESIGN:
Intervention Model Description: First, we will test the savety and effects of neuromodulation using four different tecniques on autonomous system of healthy people.
  Then, we will test the effect of neuromodulation through, vagal stimulation, on pain, fatigue, mental healthy and disautonomy of people with primary chronic pain and/or post-COVID syndrom. For this, active and sham stimulations will be compared.
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (3):
- Healthy subjects (Other): Once a week, each subject will receive a random stimulation in one of the following areas: (i) the afferent portion of the vagal nerve on the Cymba Conchae of the left ear (taVNS); (ii) rPMS on an efferent portion of the vagal nerve on the neck; (iii) rTMS intermittent theta- burst on the left DLPFC; (iv) simulated taVNS (SHAM) on helix left ear or.
  Interventions: Device: taVNS - transauricular vagal nerve stimulation; Device: rPMS - repetitive peripheric magnetic stimulation; Device: rTMS - repetitive transcranial magnetic stimulation; Device: taVNS sham
- Chronic Pain and post Covid Syndrom - Active (Experimental): These volunteers will receive 30 minutes of taVNS on the afferent portion of the vagal nerve on the ears.
  Interventions: Device: taVNS - transauricular vagal nerve stimulation
- Chronic Pain and post Covid Syndrom - Sham (Sham Comparator): These volunteers will receive 30 minutes of simulated taVNS on the afferent portion of the vagal nerve on the ears. For this, the equipment will be programmed to be on only for 1 minute.
  Interventions: Device: taVNS sham

INTERVENTIONS:
Device: taVNS - transauricular vagal nerve stimulation — 30 minutes of electrical stimulation on the afferent portion of the vagal nerve on the cymba conchae of the ear, in the following configuration: 30 seg ramp up, 30 seg on, 30 seg off in intensity on which the volunteer feels a light tingling.
  Arms: Chronic Pain and post Covid Syndrom - Active; Healthy subjects
Device: rPMS - repetitive peripheric magnetic stimulation — Magnetic stimulation on the efferent portion of the vagal nerve on the neck, on the following configuration: 20Hz, 25 pulses in the trein, in every inhalation, for 20 inhalations with 50% of machine capacity (500 pulses total).
  Arms: Healthy subjects
Device: rTMS - repetitive transcranial magnetic stimulation — rTMS intermitent theta- burst on the left DLPFC, on the following configuration: 50 Hz in treins of 5Hz, with 110% of the resting motor limiar and 600 pulses in 3 minutes.
  Arms: Healthy subjects
Device: taVNS sham — Simulated taVNS (SHAM) on helix left ear, that is the same as taVNS, but during only 1 minute
  Arms: Chronic Pain and post Covid Syndrom - Sham; Healthy subjects

SUMMARY:
The aim of this study is to analyse whether there is an advantage in adding low-intensity electrical stimulations to the vagus nerve with electrodes in the outer ear to control pain and fatigue in people with primary chronic pain, and in people who have had COVID-19. Several studies have shown that many people with primary chronic pain and also people who have had COVID patients continue to have pain and fatigue that may be due to changes that occur in the brain and the vagus nerve that passes through the neck might cause inflammation. Therefore the aim of this study is to investigate if these electrical stimulations can help improve the condition of the brain and nerve and consequently, the inflammation so that these complaints improve.

This study will be organized as the following: It will begin with an assessment, divided into a part with questionnaires and another with specific tests. The questionnaires are aimed at understanding volunteer's characteristics, pain, fatigue, inflammation, sleep, quality of life, and the presence of symptoms of anxiety and depression. Next, the volunteer will undergo two tests to assess the behavior of his/her brain. They are performed using EEG electroencephalography and transcranial magnetic stimulation (TMS).

* Quantitative EEG at rest - In this technique, a cap with electrodes is placed on volunteer's head, in contact with hair, which are connected through a gel. The volunteer needs to remain still for 6 minutes with eyes closed, sitting in a comfortable chair.
* TMS with EEG - First, the volunteer will be asked to honestly answer the questions in the safety questionnaire for using this technique. Honest answers will eliminate the risks associated with this evaluation. Next, the volunteer's skin will be cleaned with alcohol and a special paste and place three self-adhesive electrodes on the muscle of the volunteer's hand, in a muscle called the interosseous, on the side where he/she writes. These electrodes will only capture the electrical activity of the muscle. Next, a series of magnetic pulses will be administered to the volunteer's skull, in the area that controls the hand muscle. It will contract with each pulse and, with this, so that the functioning of this connection can be understood. At the same time, the EEG device will capture the brain activities that occur during this TMS stimulation. During this exam, the volunteer may feel anything from no stimulation to muscle contractions that move his/her hand. Some people also experience redness under the electrodes, fatigue, or muscle/joint pain.

After the assessments, volunteers will be randomly selected to receive neuromodulation sessions using low-intensity electrical stimulation of the vagus nerve, using electrodes in the outer ear (active group), or sessions that only simulate this neuromodulation (sham, or placebo, group). This will occur for five consecutive days, starting on the day of the assessment. This stimulation is very weak and may not even be felt by the person receiving it. This technique is safe and the most that may occur is redness or itching of the skin. A few people may also experience tingling, a burning sensation or momentary local pain, fatigue, drowsiness, difficulty concentrating and a feeling of nervousness during or after the stimulation.

At the end of the 5 days of electrical stimulation, the same initial assessments will be repeated to see if anything has changed in the volunteer's brain, heart rate, blood pressure, pain, fatigue, inflammation, sleep, quality of life, depression, and anxiety.

ELIGIBILITY:
Inclusion Criteria:

* Healthy individuals, both sexes, aged between 18 and 40 years (first arm).
* Diagnosis of primary chronic pain (for more than 3 months), such as fibromyalgia (chronic widespread pain), primary chronic headache and orofacial pain, chronic primary visceral pain, post-COVID pain, and chronic primary musculoskeletal pain;
* In the case of post-COVID-19 pain, the symptoms must be present for at least 12 weeks. The complaints of pain, fatigue, and/or changes in mental health should have started after infection by SARS-Cov-2.

Exclusion Criteria:

* Individuals who present dysautonomia;
* obese individuals with a high abdominal fat index characterized by a waist/hip ratio of 0.80 for women and 0.95 for men;
* heart disease;
* diabetes mellitus;
* vestibular alterations characterized by the Dix-Hallpike maneuver, supine rotation test, arc test, side-lying maneuver, and post-head-shake nystagmus;
* diagnosis of epilepsy or first-degree family history of epilepsy
* fever;
* chronic consumption of alcohol, or other recreational drugs;
* presence of contraindications for the use of non-invasive neuromodulation;
* those who become ill with COVID-19 during the data collection period;
* those who are unable to answer the evaluation questionnaires;
* those with clinical instability;
* those who have a previous history of chronic pain or fatigue before contracting COVID-19;
* those who have neuropathic pain.

Ages: 18 Years to 64 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 55 (Estimated)
Dates: Start 2024-04-21 (Actual); Primary Completion 2024-12-16 (Estimated); Study Completion 2024-12-16 (Estimated)

PRIMARY OUTCOMES:
Pain | 5 days
  It will be assessed through the Brief Pain Inventory (BPI), that assess place and pain intensity and its impact in life and by multidimensional pain assessment instruments to evaluate pain experience and self-efficacy

SECONDARY OUTCOMES:
Heart rate variability and blood preasure | 5 days
  It will be done using a chest polar and a sphygmomanometer.
Pressure pain threshold. | 5 days
  Assessed through handgrip dynamometry.
TMS-Evoked potential | 5 days
  TMS-Evoked Potential is a measure derived from TMS stimulus on the brain which represent a brain reactivity to exogenous stimulus
Disautonomy, fatigue and mental health | 5 days
  Dysautonomia will be assessed through TMS-EEG. Fatigue will be assessed by physical, cognitive and psychosocial fatigue scales and fatigue perception questionnaire. Mental health will be assessed by anxiety, depression and sleep quality questionnaires. Quality of life will be assessed by a specific questionnaire.

CONTACTS AND LOCATIONS:
Overall Officials: Tiago S Lopes, PhD, Study Chair — Federal University of ABC
Locations (1):
- Federal University of ABC, Sâo Bernardo Do Campo, São Paulo, Brazil

IPD SHARING:
Plan to Share IPD: No